CLINICAL TRIAL: NCT06699121
Title: A Phase 2 Randomized, Double Blind, Placebo Controlled, Parallel Study Evaluating the Safety and Efficacy of LB P8 in Patients With Primary Sclerosing Cholangitis (PSC)
Brief Title: A Study to Assess the Safety and Efficacy of LB-P8 in Patients With PSC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: LISCure Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LB08-211
Record Dates: First submitted 2024-11-17; First posted 2024-11-21 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Primary Sclerosing Cholangitis (PSC)
Keywords: PSC; Pruritus; Inflammatory bowel disease; IBD; Itch; Cholestasis
MeSH Terms: conditions — Cholangitis, Sclerosing; Pruritus; Inflammatory Bowel Diseases; Cholestasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LB-P8 low-dose (Experimental): Oral capsule, 1×10^10 CFU/day
  Interventions: Drug: LB-P8 low-dose
- LB-P8 high-dose (Experimental): Oral capsule, 1×10^11 CFU/day
  Interventions: Drug: LB-P8 high-dose
- Placebo (Placebo Comparator): Oral capsule, placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LB-P8 low-dose — One capsule QD (1×10^10 CFU/day) oral administration
  Arms: LB-P8 low-dose
Drug: LB-P8 high-dose — One capsule QD (1×10^11 CFU/day) oral administration
  Arms: LB-P8 high-dose
Drug: Placebo — One capsule QD oral administration
  Arms: Placebo

SUMMARY:
The study is designed to assess the safety and efficacy of LB-P8 in patients with primary sclerosing cholangitis.

DETAILED DESCRIPTION:
This is phase 2, randomized, double-blind, placebo-controlled, multicenter study to assess the safety and efficacy of LB-P8 in adult patients with primary sclerosing cholangitis(PSC).

* Part 1 will evaluate safety and tolerability of 2 pre-selected dose level of LB-P8 (low-dose[1×10^10 CFU/capsule] and high dose [1×10^11 CFU/capsule]) in adult patients with PSC. Part 1 plans to enroll a maximum number of 12 patients based on a "3+3" study design.
* Part 2 will evaluate safety and efficacy in adult patients with PSC. Eligible patients with PSC will be randomized in a 1:1:1 ratio to receive treatment with low-dose LB-P8(1×10^10 CFU/capsule), high-dose LB-P8(1×10^11 CFU/capsule) or matched placebo capsule. Part 2 plans to enroll and randomize 75 patients to obtain 60 evaluable patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 75 years
* A diagnosis of PSC based on cholangiographic evidence of PSC in accordance with American Association for the Study of Liver Diseases (AASLD) guidelines
* ALP >1.5 times the ULN at screening
* PSC with or without IBD, such as ulcerative colitis or Crohn's disease
* If patients are being administered biologic or advanced therapeutic treatments, immunosuppressants, systemic corticosteroids, obeticholic acid, fibrates, or statins, they must be on a stable dose for ≥3 months prior to, and including, Day 0 and plan to remain on a stable dose throughout the study
* If patients are receiving ursodeoxycholic acid, they must be on a stable dose (not exceeding 23 mg/kg/day) for >3 months prior to screening
* Patient agrees to stop all probiotics for at least 2weeks prior to treatment
* Patient is unable to conceive and/or patient who's partner is unable to become pregnant and/or agree to use effective methods of contraception when engaging in heterosexual intercourse

Exclusion Criteria:

* Treatment with any investigational agents within 3 months or 5 half-lives, whichever is longer prior to treatment or during the study. Gene therapy or other long-lasting investigational agents with unknown half-life is not allowed
* History of a liver transplant or anticipated need for a liver transplant within 1 year
* Patients who show evidence of significant worsening of hepatic function will be excluded.
* Evidence of compensated or decompensated cirrhosis based on histology, relevant medical complications, or laboratory parameters
* Model for end-stage liver disease (MELD) score as below, unless the MELD is driven by anticoagulant therapy, vitamin deficiency, or kidney disease:
* MELD Score of >12 (decompensated cirrhosis) for Part 1 of the study
* MELD Score of >12 for Part 2 of the study
* Small-duct PSC (in the absence of large duct PSC)
* Secondary causes of sclerosing cholangitis including IgG4 associated sclerosing cholangitis
* Any history of cholangiocarcinoma, gallbladder cancer, or hepatocellular carcinoma
* History of any malignancy with lymph node or regional metastases within 5 years or current malignancy undergoing active treatment
* Patients who require chronic use of antibiotics, received antibiotics in the last 1 month, or received Rebyota or Vowst (applicable for patients with Clostridioides difficile infection)
* In patients with ulcerative colitis, partial Mayo score of >6 or, patients with Crohn's disease if CDAI of >220
* Chronic kidney injury
* Recent acute cholangitis (within 90 days)
* Patients with indwelling biliary drain (or stent), total proctocolectomy with ileal anal pouch, partial large bowel resections or history of small bowel resection
* Other causes of liver disease, such as autoimmune hepatitis (AIH), primary biliary cholangitis (PBC), AIH/PSC overlap syndrome, alpha-1-antitrypsin deficiency, viral hepatitis, iron overload syndrome, Wilson disease, nonalcoholic steatohepatitis, and/or alcohol related liver disease. Additionally, positive serology for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (anti HCV) (detectable HCV RNA in the serum), or human immunodeficiency virus antibodies (anti HIV)
* Active drug (known or suspected use of illicit drugs or drugs of abuse) or alcohol abuse disorder
* Female patients who are pregnant, nursing, or planning to become pregnant during the study
* Clinically significant and/or active infection
* Subjects with a greater degree of immunosuppression, as evidenced by Alsolute neutrophil count <500 cells/mL or in the investigator's judgement immunosuppressed and at higher risk of infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of 2 different doses of LB-P8 | (Part 1) Up to 4 weeks of treatment from the Baseline
  Occurrence of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) by CTCAE V5.0
Safety and tolerability of LB-P8 | (Part 2) Up to 24 weeks of treatment from the Baseline
  Occurrence of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) by CTCAE V5.0
Mean percent change from baseline in Serum Concentrations of Alkaline Phosphatase (ALP) | (Part 2) Up to 24 weeks of treatment from the Baseline

SECONDARY OUTCOMES:
Change from baseline in ALP | (Part 2) Up to 24 weeks of treatment from the Baseline
Percentage of patients who achieve ALP of <1.5 × upper limit of normal (ULN) | (Part 2) Up to 24 weeks of treatment from the Baseline
Change from baseline in enhanced liver fibrosis (ELF™) | (Part 2) Up to 24 weeks of treatment from the Baseline
  Hyaluronic acid, procollagen-3 N-terminal peptide, and a tissue inhibitor of metalloproteinase 1 will be assessed in blood for ELF test.
Changes from baseline in biliary metrics (biliary strictures and dilatations) | (Part 2) Up to 24 weeks of treatment from the Baseline
  Biliary metrics (biliary strictures and dilatations) will be assessed by magnetic resonance cholangiopancreatography (MRCP)
Changes from baseline in liver stiffness | (Part 2) Up to 24 weeks of treatment from the Baseline
  Liver stiffness will be measured by transient elastography (FibroScan®)
Change from baseline in alanine aminotransferase (ALT) | (Part 2) Up to 24 weeks of treatment from the Baseline
Change from baseline in aspartate aminotransferase (AST) | (Part 2) Up to 24 weeks of treatment from the Baseline
Change from baseline in gamma glutamyl transferase (GGT) | (Part 2) Up to 24 weeks of treatment from the Baseline
Change from baseline in prothrombin time (PT) and partial prothrombin time (PTT) | (Part 2) Up to 24 weeks of treatment from the Baseline
Change from baseline in international normalized ratio (INR) | (Part 2) Up to 24 weeks of treatment from the Baseline
Change from baseline in total and direct bilirubin | (Part 2) Up to 24 weeks of treatment from the Baseline
Change from baseline in fasting serum bile acid level | (Part 2) Up to 24 weeks of treatment from the Baseline
The percentage of patients who experience liver disease progression | (Part 2) Up to 24 weeks of treatment from the Baseline
  The percentage of patients who experience progression to cirrhosis, clinical decompensation rates, liver transplant, newly diagnosed cholangiocarcinoma, MELD score increase from <12 to >15 and Death from any cause

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of California Davis, Sacramento, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - University Of Iowa Hospitals And Clinics, Iowa City, Iowa
  - Mercy Medical Center, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - The Vanderbilt Clinic, Nashville, Tennessee
  - Liver institute Northwest, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No